CLINICAL TRIAL: NCT06988761
Title: The Clinical Impact of Integrated Behavioral Health Techniques in Patients With Fibromyalgia: A Mayo Clinic-Lin Health Randomized Controlled Trial
Brief Title: The Clinical Impact of Integrated Behavioral Health Techniques in Patients With Fibromyalgia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elizabeth C. Wight, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-000227
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Subjects in the experimental group will receive Mayo Clinic's usual standard of care and Lin Health interventions.
  Interventions: Behavioral: Longitudinal Behavioral Health Techniques
- Control Group (Active Comparator): Subjects in control group will receive Mayo Clinic's usual standard of care.
  Interventions: Behavioral: Standard of care treatment for Fibromyalgia

INTERVENTIONS:
Behavioral: Standard of care treatment for Fibromyalgia — Patients will receive standard of care as decided by treating physician which may include patient education, physical therapy, occupational therapy, cognitive behavioral therapy, biofeedback therapy, massage, acupuncture, graded activity therapy, sleep hygiene therapy, relaxation therapies, and meditative movement therapies.
  Arms: Control Group
Behavioral: Longitudinal Behavioral Health Techniques — Patients will receive standard of care as decided by treating physician, along with the integration of longitudinal behavioral health techniques provided by Lin Health. Patients have 24/7 access to digital content and will be able to interact directly with care team members on average three times per week.
  Arms: Experimental Group

SUMMARY:
The purpose of this research is to assess the impact of using Lin Health to provide virtual long-term follow up care for patients with a diagnosis of fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must have a diagnosis of Fibromyalgia.
* Patient must be being seen at the Mayo Clinic Fibromyalgia and Chronic Fatigue Clinic in Rochester, MN.
* Patient must be able to understand and provide informed consent and HIPAA authorization
* Patient must be willing and able to complete all aspects of the study.
* Patient must be able to speak and read English.

Exclusion Criteria:

* Patient who is under the age of 18 years old.
* Patient who is unable to provide informed consent or HIPAA authorization.
* Patient who declines study participation.
* Patient who is unable to speak English.
* Patient who is on active cancer therapy.
* Patient who is actively psychotic or actively suicidal.
* Patient who is deemed inappropriate to the study by the medical professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire - Revised | Baseline, 3 months
  The Revised Fibromyalgia Impact Questionnaire (FIQR) is a self-report questionnaire designed to assess the impact of fibromyalgia on a patient's daily life. It evaluates function, overall impact, and symptoms experienced in the past 7 days. The FIQR uses an 11-point numeric scale (0 to 10) for each of the 21 questions, with higher scores indicating a greater impact of fibromyalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Wight, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No